CLINICAL TRIAL: NCT04317560
Title: Evaluation Of The Clinical Efficacy Of Liquid Platelet Rich Fibrin Application In Painful Temporomandibular Joint Disorders
Brief Title: Evaluation Of Efficacy Of Liquid Platelet Rich Fibrin In Temporomandibular Joint Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Burcu Gürsoytrak, Assistant Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-049
Record Dates: First submitted 2020-03-03; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Liquid Platelet Rich Fibrin; Temporomandibular Joint Disorders; Wilkes classification
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Arthrocentesis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthrocentesis (Active Comparator): 2 guiding points have been created on the skin. The first one is 10 mm in front of the tragus and 2 mm below the tragus line. The second guide point is on the same line, 20 mm in front of the tragus and 6 mm below. After the auriculotemporal nerve block was made, the first 20 gauge needle was inserted from the first point. 2mL Ringer's Lactate solution is injected into the temporomandibular joint area, and then a second 20 gauge needle is entered from the second guide point determined before and pressurized washing is performed with 100 mL of 5% lactate solution to enter the first needle and exit from the second needle.
  Interventions: Procedure: Arthrocentesis
- Arthrocentesis plus i-PRF injection (Experimental): 2 tubes of blood were collected from the patients with the help of vacuumed 10 mL special liquid PRF tubes (Choukroun I-PRF Collection Tubes, Dr. Choukroun) after arthrocentesis. Blood tubes were centrifuged at 700rpm for 3 minutes. 3 mL of liquid PRF was obtained at the top of each tube. Only the second needle was removed without removing the first needle inserted. I-PRF was injected into the joint areas of all patients in the experimental group, with a maximum dose of 2 mL per joint.
  Interventions: Procedure: Arthrocentesis; Procedure: injectable platelet rich fibrin injection

INTERVENTIONS:
Procedure: Arthrocentesis — 2 guiding points have been created on the skin. The first one is 10 mm in front of the tragus and 2 mm below the tragus line. The second guide point is on the same line, 20 mm in front of the tragus and 6 mm below. After the auriculotemporal nerve block was made, the first 20 gauge needle was inserted from the first point. 2mL Ringer's Lactate solution is injected into the temporomandibular joint area, and then a second 20 gauge needle is entered from the second guide point determined before and pressurized washing is performed with 100 mL of 5% lactate solution to enter the first needle and exit from the second needle.
Procedure: injectable platelet rich fibrin injection — 2 tubes of blood were collected from the patients with the help of vacuumed 10 mL special liquid PRF tubes (Choukroun I-PRF Collection Tubes, Dr. Choukroun) after arthrocentesis. Blood tubes were centrifuged at 700rpm for 3 minutes. 3 mL of liquid PRF was obtained at the top of each tube. I-PRF was injected into the joint areas of all patients in the experimental group, with a maximum dose of 2 mL per joint.
  Arms: Arthrocentesis plus i-PRF injection

SUMMARY:
This randomized clinical trial aims to evaluate the efficacy of liquid platelet-rich fibrin administration at different Wilkes stages.

DETAILED DESCRIPTION:
Thirty six patients with unilateral painful internal derangement (ID) (Wilkes' 3-4-5) were included. Patients were divided into 2 groups. In group 1 were treated with only artrosythesis. In group 2 were treated with artrosythesis and liquid platelet rich fibrin. In group 2, patients were injected with 1.5-2cc of liquid platelet-rich fibrin within the superior joint space at operation day. Pain and subjective dysfunction were recorded using a visual analog scale and Helkimo index at operation day and tenth day, one month later and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral internal temporomandibular disorder
* localized temporomandibular joint pain
* Scoring 3 and above in Wilke's classification.

Exclusion Criteria:

* Autoimmune diseases
* Significant mechanical obstruction that prevents mouth opening
* Acute capsulitis,
* Benign or malignant temporomandibular joint lesions
* Neurological disorders,
* Blood diseases and coagulation disorders
* Patients with a history of allergies or anaphylactic shock.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Helkimo Clinical Dysfunction Score improvement over time | operation time, tenth day, end of first month, end of third month
  In the Helkimo Clinical Dysfunction Index, the maximum mandibular movement limits are measured vertically and laterally. In addition, TMJ function, muscle pain, TMJ region pain and mandibular motion pain are evaluated separately. After all these evaluations, all the scores given are summed up and a total dysfunction score is obtained. If this total score is 0, the dysfunction is completely healed. If the total score is between 1 and 4, mild dysfunction, between 5 and 9, moderate dysfunction, and between 10 and 25 severe dysfunction.
  Since lower scores represent better health, the amount of improvement between sessionsis calculated by subtracting the next score from the previous score.
Visual Analog Scale improvement over time | operation time, tenth day, end of first month, end of third month
  The patient gives his pain a value between 0-10. The patients' pain scores were recorded by using a 10 cm visual analog scale (VAS) from 0, which represents no pain, to 10, which represents the worst possible pain.
  Since lower scores represent better health, the amount of improvement between sessionsis calculated by subtracting the next score from the previous score.
Maximum incisal opening improvement over time | operation time, tenth day, end of first month, end of third month
  It is the vertical distance between the incisal teeth when the patient opens his mouth to the maximum. It is measured with the help of a caliper.
  Since higher scores represent better health, the amount of improvement between sessionsis calculated by subtracting the previous score from the next score.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu GURSOYTRAK, Study Director — Aydin Adnan Menderes University
Locations (1):
- Aydın Adnan Menderes University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Albilia J DMD, MSc, Herrera-Vizcaino C DDS, Weisleder H BSc, Choukroun J MD, Ghanaati S MD, DMD, PhD. Liquid platelet-rich fibrin injections as a treatment adjunct for painful temporomandibular joints: preliminary results. Cranio. 2020 Sep;38(5):292-304. doi: 10.1080/08869634.2018.1516183. Epub 2018 Sep 20. PMID 30231809
- [Background] Pihut M, Szuta M, Ferendiuk E, Zenczak-Wieckiewicz D. Evaluation of pain regression in patients with temporomandibular dysfunction treated by intra-articular platelet-rich plasma injections: a preliminary report. Biomed Res Int. 2014;2014:132369. doi: 10.1155/2014/132369. Epub 2014 Aug 3. PMID 25157351
- [Background] Zardeneta G, Milam SB, Schmitz JP. Elution of proteins by continuous temporomandibular joint arthrocentesis. J Oral Maxillofac Surg. 1997 Jul;55(7):709-16; discussion 716-7. doi: 10.1016/s0278-2391(97)90583-8. PMID 9216503
- [Background] Helkimo M. Studies on function and dysfunction of the masticatory system. II. Index for anamnestic and clinical dysfunction and occlusal state. Sven Tandlak Tidskr. 1974 Mar;67(2):101-21. No abstract available. PMID 4524733
- [Background] Nitzan DW, Samson B, Better H. Long-term outcome of arthrocentesis for sudden-onset, persistent, severe closed lock of the temporomandibular joint. J Oral Maxillofac Surg. 1997 Feb;55(2):151-7; discussion 157-8. doi: 10.1016/s0278-2391(97)90233-0. PMID 9024352